CLINICAL TRIAL: NCT01288547
Title: Temporal Change of Mood and Cognition in Healthy Subjects After Consumption of Theobromine and/ or Caffeine
Brief Title: Effects of Theobromine and Caffeine on Mood, Cognition and Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unilever R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 07045V
Record Dates: First submitted 2011-01-31; First posted 2011-02-02 (Estimated); Last update posted 2012-02-23 (Estimated); Status verified 2012-02

CONDITIONS: Mood
Keywords: cognition; attention; methylxanthine
MeSH Terms: interventions — Theobromine; Caffeine; methylxanthine; Cellulose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- theobromine (Active Comparator): theobromine (700 mg) in capsule
  Interventions: Dietary Supplement: theobromine
- caffeine (Active Comparator): caffeine (120 mg) in capsule
  Interventions: Dietary Supplement: Caffeine
- Placebo capsule (Placebo Comparator): no theobromine or caffeine
  Interventions: Dietary Supplement: placebo
- theobromine + caffeine (Active Comparator): Combined theobromine and caffeine treatment, consisting of 700 mg theobromine and 120 mg caffeine
  Interventions: Dietary Supplement: caffeine + theobromine

INTERVENTIONS:
Dietary Supplement: theobromine — 700 mg theobromine in gelatin capsules given one time only
  Other Names: 3,7-dimethylxanthine
  Arms: theobromine
Dietary Supplement: Caffeine — 120 mg caffeine in capsules given one time only
  Other Names: 1,3,7-trimethylxanthine
  Arms: caffeine
Dietary Supplement: caffeine + theobromine — 120 mg caffeine and 700 mg theobromine in capsules given one time only
  Other Names: methylxanthines
  Arms: theobromine + caffeine
Dietary Supplement: placebo — cellulose in capsules given one time only
  Other Names: avicel (cellulose)
  Arms: Placebo capsule

SUMMARY:
The purpose of this study was to measure potential mood, cognition and blood pressure effects of theobromine and caffeine in healthy women

DETAILED DESCRIPTION:
Background Previous research has shown that naturally occurring chocolate ingredients theobromine and caffeine have positive effects on mood.

Objectives: To assess mood and cognition in adult subjects after the consumption of capsules filled with 1. placebo, 2. theobromine alone, 3. caffeine alone or, 4. theobromine and caffeine combined together.

Study design: Double-blind, placebo-controlled, randomized, cross-over design, with a 1 week washout period in between.

During the 4 weeks intervention period, once a week one of the 4 types of test products were consumed with 250ml of water in a randomized order;

1. placebo capsules
2. theobromine capsules (700 mg),
3. caffeine capsules (120 mg),
4. mix of theobromine (700 mg) and caffeine (120 mg). Twenty-four healthy female subjects (and 4 reserve subjects) were recruited for a four week intervention period in total with every week a 4 hrs measurement day and one of the interventions.

Primary parameters: mood (via a Bond-Lader/ caffeine visual analogue questionnaire), cognition (Digit Symbol substitution) Secondary parameters: blood pressure

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age at start of study 18 till 70 years
* Body Mass Index (BMI) between 20 and 30 kg/m2 inclusive
* Reported alcohol consumption for females < 21
* Willing to refrain from caffeine and theobromine for 24 hours
* Apparently healthy: no reported current or previous metabolic diseases, chronic gastrointestinal disorders, cardiovascular or psychiatric disease which might effect study measurements assessed by Research physician
* willing to consume animal foods products (gelatine).
* Consumes caffeine (7 cups of either tea, cola or coffee per week minimum)
* Having a general practitioner (GP)

Exclusion Criteria:

* Being an Unilever employee
* Blood pressure above 160/90 mmHg at screening and irregular heart rate
* Using or planning to use any medically prescribed diet or weight-loss diet
* Reported intense sporting activities > 10 h/w
* Subjects who undergoing medical treatment that may interfere with the study outcome.
* Reported weight change ± 10% during a period of 6 months prior to the study
* Reported intolerance or allergy for one of test products or standardized meal
* The habit of smoking during the past half year, drug use during the past half year or using nicotine containing medicines during the past month
* Reported lactating (or lactating < 6 weeks ago), pregnant (or pregnant < 3 months ago) or wish to become pregnant during the study
* Not able to perform the computer tasks assessed during screening
* Reported participation in night shift work during the study period

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-05; Primary Completion 2008-06 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Mood and cognition | 3 hrs every week for 4 weeks
  Bond Lader Visual Analogue Scale
  Digit Symbol Substitution
  Caffeine Negative Symptoms

SECONDARY OUTCOMES:
blood pressure and heart rate | 3 hrs every week for 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Zebregs, Principal Investigator — Unilever R&D
Locations (1):
- Unilever Discover, Vlaardingen, South Holland, Netherlands